CLINICAL TRIAL: NCT00119873
Title: A Phase I Dose-Escalation Clinical Trial to Evaluate the Safety and Immunogenicity of a Multiclade, Multivalent Recombinant Adenoviral Vector HIV Vaccine, VRC-HIVADV014-00-VP, in Healthy, HIV-1 Uninfected Adult Participants Who Have Low Titers of Pre-Existing Ad5 Neutralizing Antibodies
Brief Title: Safety of and Immune Response to an Experimental HIV Vaccine (VRC-HIVADV014-00-VP) in HIV Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 054; 10121 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2005-07-12; First posted 2005-07-14 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Preventive Vaccine; AIDS Vaccines; Adenoviridae
MeSH Terms: conditions — HIV Infections; Adenoviridae Infections

INTERVENTIONS:
Biological: VRC-HIVADV014-00-VP

SUMMARY:
The purpose of this study is to determine the safety of and immune response to an experimental HIV vaccine in HIV uninfected individuals.

DETAILED DESCRIPTION:
The HIV epidemic is a major global health challenge. People in developing nations have limited access to life-sustaining antiretrovirals and account for over 95% of the 5 million new HIV infections annually. The development of a safe, effective, and widely accessible HIV vaccine is paramount in these areas. The adenoviral vector vaccine VRC-HIVADV014-00-VP has been shown to elicit a CD8 cytotoxic lymphocyte (CTL) response believed to be crucial in an effective preventive HIV vaccine. The purpose of this study is to determine the safety and immunogenicity of VRC-HIVADV014-00-VP in HIV uninfected adults. In this study, HIV uninfected individuals with low levels of pre-existing adenovirus neutralizing antibodies will receive different doses of the preventive vaccine to determine its safety, tolerability, and immunogenicity.

This study will last 1 year. Participants will be randomly assigned to one of two groups. At study entry, participants in each group will receive a single injection of either one of two doses of the adenoviral vector vaccine or placebo. Participants will record their temperature and other side effects in a symptom log on the day of vaccination and for 3 days thereafter. Participants will have seven clinic visits over 12 months. A physical exam, HIV and pregnancy prevention counseling, and blood and urine collection will occur at each visit. Participants will also be asked about side effects they may be experiencing and medications they are taking.

ELIGIBILITY:
Inclusion Criteria:

* Have access to a participating site and are willing to be followed for the duration of the study
* Willing to receive HIV test results
* Able to understand and comply with study requirements
* In good general health
* Have neutralizing adenovirus antibody levels that are less than a 1:12 ratio
* Agree to use acceptable methods of contraception for at least 21 days prior to study start and for the duration of the study.

Exclusion Criteria:

* HIV infected
* Positive hepatitis B surface antigen
* Positive anti-hepatitis C virus antibodies
* Prior receipt of an HIV vaccine
* Immunosuppressive drugs within 168 days prior to first vaccination
* Have received donated blood within 120 days prior to first vaccination
* Have received immunoglobulin within 60 days of the first vaccination
* Live attenuated vaccines or investigational research agents within 30 days prior to first vaccination
* Subunit or killed vaccines within 14 days prior to first vaccination
* Current preventive or therapeutic anti-tuberculosis (TB) treatment
* Any medical, psychiatric, or social condition that would interfere with the study
* Any occupational or other responsibility that would interfere with the study
* Serious adverse reactions to vaccines
* Autoimmune disease
* Immunodeficiency
* Active syphilis infection. Participants who have been fully treated for syphilis over 6 months prior to study entry are not excluded.
* Asthma. Participants who have had completely resolved childhood asthma are not excluded.
* Diabetes mellitus type I or II. Participants who have had isolated gestational diabetes are not excluded.
* Thyroid disease or removal of the thyroid
* Blood vessel swelling within the last 3 years
* Uncontrolled hypertension
* Body mass index (BMI) of 40 or higher
* Bleeding disorder
* Cancer. Participants whose cancer has been removed and is unlikely to recur during the study are not excluded.
* Seizure disorder. Participants who have not required medication or had a seizure for 3 years prior to study entry are not excluded.
* Removal of the spleen or have a nonfunctioning spleen
* Psychiatric conditions that may interfere with the study
* Pregnancy, breastfeeding, or plan to become pregnant during the study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Blood and chemical parameters for 12 months after injection
Local and systemic adverse reactions for 12 months after injection

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Peiperl, MD, Study Chair — San Francisco Department of Public Health
Locations (3):
- United States (3):
  - San Francisco Vaccine and Prevention CRS, San Francisco, California
  - Vanderbilt Vaccine CRS, Nashville, Tennessee
  - FHCRC/UW Vaccine CRS, Seattle, Washington

REFERENCES:
- [Background] Shiver J. A non-replicating adenoviral vector as a potential HIV vaccine. Res Initiat Treat Action. 2003 Spring;8(2):14-6. PMID 12845771
- [Background] Casimiro DR, Bett AJ, Fu TM, Davies ME, Tang A, Wilson KA, Chen M, Long R, McKelvey T, Chastain M, Gurunathan S, Tartaglia J, Emini EA, Shiver J. Heterologous human immunodeficiency virus type 1 priming-boosting immunization strategies involving replication-defective adenovirus and poxvirus vaccine vectors. J Virol. 2004 Oct;78(20):11434-8. doi: 10.1128/JVI.78.20.11434-11438.2004. PMID 15452269
- [Background] Shiver JW, Emini EA. Recent advances in the development of HIV-1 vaccines using replication-incompetent adenovirus vectors. Annu Rev Med. 2004;55:355-72. doi: 10.1146/annurev.med.55.091902.104344. PMID 14746526
- [Background] Gomez-Roman VR, Robert-Guroff M. Adenoviruses as vectors for HIV vaccines. AIDS Rev. 2003 Jul-Sep;5(3):178-85. PMID 14598567
- [Result] Peiperl L, Morgan C, Moodie Z, Li H, Russell N, Graham BS, Tomaras GD, De Rosa SC, McElrath MJ; NIAID HIV Vaccine Trials Network. Safety and immunogenicity of a replication-defective adenovirus type 5 HIV vaccine in Ad5-seronegative persons: a randomized clinical trial (HVTN 054). PLoS One. 2010 Oct 27;5(10):e13579. doi: 10.1371/journal.pone.0013579. PMID 21048953